CLINICAL TRIAL: NCT02093013
Title: Impact of an Integrated Care Intervention Program on Asthmatic Patients.
Brief Title: Effectiveness of an Integrated Care Program on Asthma Control and Inhaled Corticosteroids Adherence
Acronym: RESPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Line Guénette, Co-investigator, Laval University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DR-002-1077
Record Dates: First submitted 2014-03-18; First posted 2014-03-20 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Asthma
Keywords: asthma; intervention; medication adherence; inhaled corticosteroids; asthma control; integrated care
MeSH Terms: conditions — Asthma; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrated care program (Experimental)
  Interventions: Other: Integrated care program
- Control group (No Intervention): This group kept receiving usual care from their health care professionals.

INTERVENTIONS:
Other: Integrated care program — Integrated care program meant in effect, calling on the family medicine group (FMG) nurses to evaluate and support asthmatic patients. The FMG and asthma education centre (AEC) nurses received special training and followed a protocol based on the theoretical model and the Canadian asthma management recommendations then in force. The protocol had five main aspects: 1) asthma assessment, 2) self-management, 3) environment and lifestyle, 4) collaborative care plan, and 5) information sharing and follow-up.
  Arms: Integrated care program

SUMMARY:
The investigators propose to implement and evaluate an integrated care program for enhancing the care of patients with asthma in a region of Quebec province, Canada. The investigators will implement our intervention in a family medicine group practice setting and plan to deliver it to 150 experimental group subjects. The investigators will simultaneously study 300 control subjects who are receiving usual care in other regions of the province of Quebec. Our hypothesis is that the program will improve the quality of life of patients with asthma exposed to the program, asthma control, inhaled corticosteroid adherence, knowledge of asthma, and a number of variables that relate to the conceptual model selected as a framework for this study (the PRECEDE-PROCEED model of Green and Kreuter).

ELIGIBILITY:
Inclusion Criteria:

Individuals aged 12 to 45 years, for whom the pharmacists had dispensed at least one anti-asthma drug in the previous six months were screened and randomly contacted by phone. Those who reported an asthma diagnosis and who were using a short-acting beta-2-agonist (SABA) >3 times a week (except before exercise) or a corticosteroid (inhaled or oral), irrespective of frequency were included.

Exclusion Criteria:

Pregnancy, no prior asthma diagnosis, participation in an ongoing respiratory study, or another respiratory illness.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 349 (Actual)
Dates: Start 2004-05; Primary Completion 2007-01 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Asthma control | One year
  The primary outcome was asthma control, measured with the validated Asthma Control Questionnaire.

SECONDARY OUTCOMES:
Adherence to ICS | One year
  Adherence to medication for each participant reporting an inhaled corticosteroids (ICS) prescription was assessed using two measures; the validated Morisky medication adherence scale (MMAS-4) composed of 4 questions (yes/no) about past medication use patterns, and the medication possession ratio (MPR), a validated objective measure based on pharmacy records.

OTHER OUTCOMES:
Implementation of the program | One year

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyne Moisan, Ph.D., Principal Investigator — URESP, Centre hospitalier affilié universitaire de Québec
Locations (1):
- Centre hospitalier affilié universitaire de Québec, Québec, Quebec, Canada

REFERENCES:
- [Result] Jobin MS, Moisan J, Bolduc Y, Dorval E, Boulet LP, Gregoire JP. Factors associated with the appropriate use of asthma drugs. Can Respir J. 2011 Mar-Apr;18(2):97-104. doi: 10.1155/2011/426528. PMID 21499595
- [Result] Guenette L, Breton MC, Gregoire JP, Jobin MS, Bolduc Y, Boulet LP, Dorval E, Moisan J. Effectiveness of an asthma integrated care program on asthma control and adherence to inhaled corticosteroids. J Asthma. 2015;52(6):638-45. doi: 10.3109/02770903.2014.999084. PMID 25539138
- [Derived] Adouni Lawani M, Zongo F, Breton MC, Moisan J, Gregoire JP, Dorval E, Boulet LP, Jobin MS, Guenette L. Factors associated with adherence to asthma treatment with inhaled corticosteroids: A cross-sectional exploratory study. J Asthma. 2018 Mar;55(3):318-329. doi: 10.1080/02770903.2017.1326131. Epub 2017 May 26. PMID 28471286